CLINICAL TRIAL: NCT02763137
Title: A Phase IIa Study to Assess the Safety, Tolerability, Plasma Pharmacokinetics and Efficacy of Intermittent Oral Administration of Standard Levodopa/Carbidopa vs. Semi-continuous Intra-oral Administration of Levodopa/Carbidopa in Patients With Advanced Parkinson's Disease Who Suffer Motor Fluctuations
Brief Title: Intermittent Oral Administration vs. Semi-continuous Intra-oral Administration of Levodopa/Carbidopa in Fluctuating Parkinsonian Patients
Acronym: LDCD-001
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: IRCCS San Raffaele Roma (Other)
Collaborators: SynAgile Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RP 12/14
Record Dates: First submitted 2016-04-26; First posted 2016-05-05 (Estimated); Last update posted 2024-04-10 (Actual); Status verified 2022-10

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — carbidopa, levodopa drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard LD/CD (Active Comparator): Standard LD/CD administered at patient's usual dose and frequency
  Interventions: Drug: Standard LD/CD
- Semi continuous intra-oral administration of LD/CD (Experimental): Semi continuous intra-oral administration of LD/CD at a dose equivalent to the patient's regular dose of standard LD/CD
  Interventions: Drug: Semi continuous intra-oral administration of LD/CD

INTERVENTIONS:
Drug: Standard LD/CD — LD/CD will be administered at patient's usual dose and frequency during 8 hours interval
  Other Names: Sinemet 25 mg/100 mg at patient's usual dose and frequency
  Arms: Standard LD/CD
Drug: Semi continuous intra-oral administration of LD/CD — Semi continuous intra-oral administration of standard LD/CD at a dose equal to the total dose of standard oral LD/CD that patients would normally consume over 8 hours period.
  Other Names: Sinemet 25 mg/100 mg administered at 5-10 minutes intervals
  Arms: Semi continuous intra-oral administration of LD/CD

SUMMARY:
This is a phase IIa study to assess the safety, tolerability, plasma pharmacokinetics and efficacy of intermittent oral administration of standard levodopa/carbidopa (LD/CD) vs.semi-continuous intra-oral administration of levodopa/carbidopa in patients with advanced Parkinson's disease (PD) who suffer motor fluctuations.The objective of this study is to assess the plasma pharmacokinetics (PK) of continuous intra-oral administration of LD/CD vs. intermittent administration of standard oral LD/CD. For purposes of this study continuous intra-oral administration of LD/CD is defined as oral administration of LD/CD at 5-10 minute intervals.

Secondary objectives are to assess the safety and tolerability of continuous intra-oral administration of LD/CD and the effect on PD motor function of continuous intra-oral administration of LD/CD vs. intermittent administration of standard oral LD/CD.

DETAILED DESCRIPTION:
18 PD subjects with motor fluctuations on stable doses of standard levodopa/carbidopa +/- other dopaminergic therapy who meet entry criteria and sign an Institutional Ethical Committee approved informed consent will participate in this study. The study will be conducted at the San Raffaele IRCCS in Rome, Italy.

Subjects who successfully complete the screening activities to confirm eligibility and are approved by an enrollment steering committee will be admitted to hospital on the evening of day 1 to undergo baseline evaluations. Standard oral levodopa/carbidopa (LD/CD) medication will be stopped at midnight. On day 2, a standardized low protein breakfast will be provided and treatment will be initiated with their usual dose of standard oral LD/CD. All subsequent doses will be administered at their pre-baseline dosing intervals; other anti-parkinson medications will not be stopped and will be maintained at their usual dose. If rescue therapy is required, treatment with apomorphine sc will be administered as a first preference. Plasma levels of levodopa and metabolites will be measured over the course of the ensuing 8 hours. Physicians will assess motor status (off, on without dyskinesia, or on with dyskinesia) at 30-minute intervals throughout the 8-hour observation period and perform UPDRS motor exams at 0, 2, 4, and 8 hours. Patients will then resume their standard oral LD/CD anti-parkinsonian medications (if any), which will be stopped at midnight. On day 3 subjects will receive continuous intra-oral administration of standard LD/CD at a dose equal to the total dose of standard oral LD/CD that they would normally consume over the time course of the study period. For the purposes of this study continuous intra-oral administration will refer to oral dosing at 5-10 minute intervals. To achieve this, the drug will be chopped and administered with water so that the same total dose of levodopa that would normally be taken intermittently will be divided up and administered as small doses at 5-10 minute intervals. Patients will undergo all of the same PK blood sampling as on Day 2. If the patient is taking Stalevo, a dose of entacapone will be administered at the usual time intervals that Stalevo otherwise would have been taken. Patients will then resume their standard oral LD/CD anti-parkinsonian medication (if any), which will be stopped at midnight. On Day 4 of the study subjects will receive their first LD/CD dose orally, and the balance of the total dose they would normally take over the next 8 hours by way of continuous intra-oral administration of LD/CD over the course of the 8 hour study period. If taking Stalevo, entacapone will be administered by itself at the time Stalevo would normally have been taken.

Physicians will assess motor status (off, on without dyskinesia, or on with dyskinesia) at 30-minute intervals throughout the continuous intra-oral administration and perform UPDRS motor exams at 0, 2, 4, and 8 hours. At the completion of the study, patients will be discharged from the clinic on their standard medication. Patients will return on day 18 for a safety evaluation.

ELIGIBILITY:
Inclusion criteria

1. PD diagnosis consistent with United Kingdom Brain Bank Criteria
2. Good response to levodopa with at least 2 hours of wearing off episodes in judgment of investigator
3. Stable doses of levodopa plus/minus other dopaminergic therapy (minimum of 4 weeks for each drug)
4. Mini Mental Score Examination (MMSE): score > 26
5. Capable of providing informed consent
6. No clinically significant medical, psychiatric or laboratory abnormalities in the judgment of the investigator.
7. No history of psychosis or hallucinations in the past 6 months
8. Women who are capable of child bearing must have a negative urine pregnancy test at screening visit and use an adequate contraceptive method throughout the study.
9. Approval for entry into the study by an enrolment steering committee

Exclusion criteria

1. Atypical or secondary parkinsonism
2. Severe dyskinesia that might interfere with study performance in judgment of investigator
3. Patient receiving duodopa, apomorphine infusion or Deep Brain Stimulation (DBS)
4. Dysphagia or sialorrhea that might interfere with administration of study intervention
5. Any relevant medical, surgical, or psychiatric condition, laboratory value, or concomitant medication which, in the opinion of the Investigator, would interfere with performing a pharmacokinetic study or would interfere with drug absorption.

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2014-07-30 (Actual); Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Variability in the observed plasma concentration of levodopa as assessed with the fluctuation index (Fluctuation index= (Maximum Plasma Concentration (Cmax)-Minimum Plasma Concentration (Cmin))/Concentration average) | Change in fluctuation index between Day 2 and Day 3
  Change in fluctuation index between intermittent administration (Day 2) and intra-oral administration (Day 3)

SECONDARY OUTCOMES:
Assess the safety and tolerability of continuous intra-oral administration of LD/CD: Adverse Events | From Day 1 to Day 18
  Record of any adverse event
Assess the effect on number of hours of "off" time of continuous intra-oral administration of LD/CD vs. intermittent administration of standard oral LD/CD | Change in number of hours of "off" time between Day 2 and Day 3
Assess the effect on UPDRS of continuous intra-oral administration of LD/CD vs. intermittent administration of standard oral LD/CD | Change in UPDRS between Day 2 and Day 3

CONTACTS AND LOCATIONS:
Overall Officials: FABRIZIO STOCCHI, PROFESSOR, Principal Investigator — IRCCS San Raffaele
Locations (1):
- Irccs San Raffaele Pisana, Rome, Italy

IPD SHARING:
Plan to Share IPD: Yes
Publication on peer-reviewed journal

REFERENCES:
- [Result] Stocchi F, Vacca L, Ruggieri S, Olanow CW. Intermittent vs continuous levodopa administration in patients with advanced Parkinson disease: a clinical and pharmacokinetic study. Arch Neurol. 2005 Jun;62(6):905-10. doi: 10.1001/archneur.62.6.905. PMID 15956161